CLINICAL TRIAL: NCT00789503
Title: Long-Term Effects of Giving Nursing-Home Residents Bread Fortified With 125 Micrograms (5000 IU) Vitamin D3 Per Daily Serving
Brief Title: Nursing-Home Residents Given Bread Fortified With Vitamin D3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Natural Ovens of Manitowoc, Manitowoc, USA (Unknown)
Responsible Party: Dr Reinhold Vieth, Mount Sinai Hospital, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bread Vitamin D
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Vitamin D Deficiency; Low Bone Density
Keywords: dietary fortification; Vitamin D3; Osteomalacia; bread; bone mineral density; geriatrics; cholecalciferol; calcidiol; osteoporosis; dual-energy photon absorptiometry; bread fortification
MeSH Terms: conditions — Vitamin D Deficiency; Bone Diseases, Metabolic; Osteomalacia; Osteoporosis | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bread fortified with vitamin D3 and calcium (Experimental)
  Interventions: Dietary Supplement: Bread fortified with vitamin D3 and calcium

INTERVENTIONS:
Dietary Supplement: Bread fortified with vitamin D3 and calcium — Bread fortified with vitamin D3 (5000 IU per bun) and calcium

SUMMARY:
Background. For older adults, serum 25-hydroxyvitamin D (25(OH)D) higher than 75 nmol/L lowers fracture risk and attainment of this 25(OH)D target may require 125 mcg (5000 IU)/d of vitamin D3.

Objective: We wanted to characterize the safety and efficacy of fortifying bread with a biologically meaningful amount of vitamin D3.

DETAILED DESCRIPTION:
Methods: In a single-arm design, 45 nursing-home residents consumed one bun/d that had been fortified with 125 mcg (5,000 IU) of vitamin D3 and 320 mg elemental calcium.

ELIGIBILITY:
Inclusion Criteria:

* Healthy seniors in an institution in Romania

Exclusion Criteria:

* Known hypercalcemic or hypercalciuric disease

Ages: 58 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D response | 12 months

SECONDARY OUTCOMES:
Effects on serum calcium | 12 months
Effects on urine calcium | 12 months
Change in spine and hip bone mineral density, baseline vs final | 12 months
Change in parathyroid hormone, baseline vs final | 12 months

REFERENCES:
- [Derived] Mocanu V, Vieth R. Three-year follow-up of serum 25-hydroxyvitamin D, parathyroid hormone, and bone mineral density in nursing home residents who had received 12 months of daily bread fortification with 125 mug of vitamin D(3). Nutr J. 2013 Oct 11;12:137. doi: 10.1186/1475-2891-12-137. PMID 24120120
- [Derived] Mocanu V, Stitt PA, Costan AR, Voroniuc O, Zbranca E, Luca V, Vieth R. Long-term effects of giving nursing home residents bread fortified with 125 microg (5000 IU) vitamin D(3) per daily serving. Am J Clin Nutr. 2009 Apr;89(4):1132-7. doi: 10.3945/ajcn.2008.26890. Epub 2009 Feb 25. PMID 19244376